CLINICAL TRIAL: NCT04950530
Title: The Effect of Biktarvy (B/F/TAF) on Whole-body Insulin Sensitivity, Lipid and Endocrine Profile in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRF007
Record Dates: First submitted 2021-06-24; First posted 2021-07-06 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: HIV-1-infection
Keywords: HIV; Insulin; Biktarvy
MeSH Terms: conditions — Insulin Resistance | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; bictegravir

STUDY DESIGN:
Intervention Model Description: Subjects will be randomised to start on Biktarvy tablet once daily OR no treatment for the first 28 day dosing phase of the study then will cross over to the alternative for the second dosing phase, following a 2 week washout period (equivalent to 5+ B/F/TAF elimination half-lives).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Biktarvy - one tablet once daily, orally administered for the first 28 days of the study.
  No treatment for the last 44 days of the study.
  Interventions: Drug: BIKTARVY 50Mg-200Mg-25Mg Tablet
- Arm 2 (Experimental): No treatment for the first 28 days of the study. Biktarvy - one tablet once daily, orally administered for the last 28 days of the study (day 44-72).
  Interventions: Drug: BIKTARVY 50Mg-200Mg-25Mg Tablet

INTERVENTIONS:
Drug: BIKTARVY 50Mg-200Mg-25Mg Tablet — A three-drug fixed dose combination tablet containing 50mg of bictegravir, 200mg of emtricitabine, and 25mg of tenofovir alafenamide taken once daily, orally
  Other Names: BIC/FTC/TAF; Bictegravir

SUMMARY:
This study will investigate changes in insulin sensitivity, lipid metabolism and endocrine profile in HIV-negative subjects exposed to Biktarvy (B/F/TAF) compared to subject not exposed to B/F/TAF for 28 days.

DETAILED DESCRIPTION:
A randomised, crossover study investigating the difference in changes in insulin sensitivity (determined by peripheral glucose uptake using a euglycaemic clamp) with the administration of Biktarvy (B/F/TAF) compared to no B/F/TAF for 28 days in HIV seronegative healthy volunteers.

Group 1:

B/F/TAF tablet once daily for the first 28 days of the study. No treatment for the last 44 days of the study.

Group 2:

No treatment for the first 28 days of the study. B/F/TAF tablet once daily for the last 28 days of the study (day 44-72).

Research bloods, endocrine profiles, weight and urine samples will be collected at baseline, as well as day 28, 44, and 72 to enable comparative analyses.

Participants will be closely monitored whilst taking the study medications. Participants will exit the study 72 days post-randomisation, with a follow-up call 28 days after exiting.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Cis-Male and Cis-Female healthy subjects without underlying conditions
* Cis-Male and Cis-Female subjects with recruitment stratified to include at least 6 female subjects and at least 6 subjects of black Africa origin
* Subjects must have documented negative HIV serology by ELISA and P24 antigen and not receiving anti-HIV pre-exposure prophylaxis (PreP)
* Subjects must be clinically well volunteers aged between 18 to 60 years with BMI <30 kg/m2 but >18 kg/m2
* Healthy, as determined by the investigator or medically qualified designee based on a medical evaluation, including medical history, physical examination, laboratory tests, and cardiac evaluation (including ECG)
* Non-fasting blood glucose, total cholesterol and triglycerides within normal limits
* Subjects should have complete blood count (FBC) with normal differential and platelet count
* A female, may be eligible to enter and participate in the study if she:

  * is of non-child-bearing potential defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy or,
  * is of child-bearing potential with a negative pregnancy test at both Screening and Day 1 and agrees to use one of the following methods of contraception to avoid pregnancy:
  * Complete abstinence from penile-vaginal intercourse. Abstinence is acceptable only as true abstinence when this is in line with the preferred and usual lifestyle of the participant;
  * Any intrauterine device with published data showing that the expected failure rate is <1% per year (not all intrauterine devices meet this criterion, see Appendix 6] for an example listing of approved intrauterine devices);
  * Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject;
  * Approved hormonal contraception (see Appendix 6] for a listing of examples of approved hormonal contraception)*;
  * Any other method with published data showing that the expected failure rate is <1% per year
* Men who have partners who are women of childbearing potential (WOCBP - definition in Appendix 6) must be using an adequate method of contraception to avoid pregnancy in their partner throughout the study and for a period of at least 4 weeks after the study;
* Complete abstinence from penile-vaginal intercourse. Abstinence is acceptable only as true abstinence when this is in line with the preferred and usual lifestyle of the patient;
* Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
* Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion, see Appendix 4 for an example listing of approved IUDs) plus male condom;
* Sterilisation confirmed prior to the subject's entry into the study
* Approved hormonal contraception used by female partner (see protocol appendix 4 for a listing of examples of approved hormonal contraception) plus male condom;
* Any other method with published data showing that the expected failure rate is <1% per year and not containing hormones plus male condom.
* Any contraception method must be used consistently, in accordance with the approved product label and for at least four weeks after discontinuation of IMP (Appendix 6).

Any contraception method must be used consistently, in accordance with the approved product label and for at least 28 days prior to the first dose of study medication and 4 weeks after discontinuing the study medication.

Exclusion Criteria:

* Subjects with a waist hip ratio > 0.97 or BMI > 30kg/m2 and BMI <18 kg/m2 will be excluded
* Acute or chronic hepatitis B infection (determined by positive hepatitis B surface antigen result at the screening visit)
* Acute or chronic hepatitis C infection (determined by positive hepatitis C antibody result at the screening visit)
* Diabetes mellitus, other metabolic syndrome or disease process in the opinion of the investigator likely to cause marked disturbance in glucose and lipid homeostasis including hypertension. Subject with HbA1c >42 mmol/mol will be excluded.
* History or presence of allergy to the B/F/TAF
* ALT greater than or equal to 1.5 x ULN and total bilirubin greater than or equal to 1.5 x ULN excluded;
* Pregnancy and breastfeeding women
* Alcohol consumption >10 units/week
* Clinically relevant drug use (positive urine drug screen) or history of alcohol or drug use considered by the Investigator to be sufficient to hinder compliance with treatment, follow-up procedures or evaluation of adverse events. Smoking is permitted, but tobacco intake should remain consistent throughout the study.
* Unable to refrain from the use of prescription (e.g., dofetilide) or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives prior to the baseline visit and throughout the study until the follow-up period, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise participant safety.
* This includes on-going therapy with any of the following

  * Metabolically active medications
  * Any lipid-lowering medication
  * Hormonal agents (oestrogens or androgens)
  * Glucocorticoids including inhaled steroids except for 'as necessary' use
  * Beta-blockers
  * Thiazide diuretics and indapamide
  * Thyroid preparations
  * Psychotropic agents
  * Anabolic steroids
  * Megestrol acetate
  * Dofetilide (or pilsicainide)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity in participants from baseline to end of study between two crossover groups | Baseline, day 28, 44, and 72 for both groups
  Change in insulin sensitivity will be determined by peripheral glucose uptake using a euglycaemic clamp.

SECONDARY OUTCOMES:
Effect of Biktarvy on adipocytokines | Baseline, day 28, 44, and 72 for both groups
  Fasting adiponectin and leptin levels in blood.
Effect of Biktarvy on fasting ghrelin | Baseline, day 28, 44, and 72 for both groups
  Fasting ghrelin levels in blood.
Effect of Biktarvy on pituitary hormones | Baseline, day 28, 44, and 72 for both groups
  Pituitary hormone function tests to measure blood levels of the following:
  Adrenocorticotrophic hormone (ACTH) Thyroid-stimulating hormone (TSH) Luteinising hormone (LH) Follicle-stimulating hormone (FSH) Prolactin (PRL) Melanocyte-stimulating hormone (MSH) Cortisol Insulin-like growth factors (IGFs)
Effect of Biktarvy on lipid profile including lipid fractions | Baseline, day 28, 44, and 72 for both groups
  Lipid profile in serum samples to measure blood levels of:
  Fasting cholesterol Triglycerides High-density lipoproteins (HDL) Low-density lipoproteins (LDL)
Effect of Biktarvy on changes in indirect calorimetry | Baseline, day 28, 44, and 72 for both groups
  Indirect calorimetry by ventilated hood expires gas analysis will be used to determine energy expenditure during the course of the clamp procedures.
Effect of Biktarvy on changes in food intake | Baseline, day 28, 44, and 72 for both groups
  Changes measured food diaries completed 3 days prior to each trial visit.
Effect of Biktarvy on quality of sleep | Baseline, day 28, 44, and 72 for both groups
  Changes measured through the Pittsburgh Sleep Quality Index (PSQI).
  Questionnaire score ranges 0-21, with higher score indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Milinkovic, Principal Investigator — Chelsea and Westminster Hospital
Locations (1):
- Chelsea & Westminster Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No